CLINICAL TRIAL: NCT04442711
Title: Pulmonary Fibrosis Biomarkers During Exacerbation
Brief Title: Cohort of IPF Patients Experiencing an Exacerbation
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Nils Hoyer, Principal Investigator, University Hospital, Gentofte, Copenhagen
Other Study IDs: PFBIO-EXA
Record Dates: First submitted 2020-06-13; First posted 2020-06-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Exacerbation; Hospitalization; Biomarkers; Outcome; Prognosis; Diagnosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum and plasma are collected within 24 hrs of hospital admission for measurement of biomarkers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PFBIO-EXA: All patients recruited for PFBIO-EXA from the original PFBIO cohort are included into the cohort.

SUMMARY:
Extension of the PFBIO cohort which includes patients with newly diagnosed idiopathic pulmonary fibrosis (IPF) for longitudinal follow-up for up to 5 years.

In the PFBIO-EXA extension, patients are included if they experience an exacerbation, or other increase in respiratory symptoms requiring hospital admission, for further collection of clinical and biological data.

DETAILED DESCRIPTION:
The aim of this study is to investigate the diagnostic and prognostic value of clinical and blood biomarkers during exacerbations, or other increase in respiratory symptoms requiring hospital admission in patients with IPF.

Patients that are already included in the PFBIO-cohort (NCT02755441) and who are admitted to hospital with an increase in respiratory symptoms, are also included in PFBIO-EXA.

Patients are recruited within 24 hrs. from hospital admission with respiratory worsening, where clinical data, and blood samples are collected. The blood samples are investigated for the same blood biomarkers as PFBIO.

Patient related outcomes are also collected, including quality-of-life questionnaires and outcomes of the exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Admitted with an increase in respiratory symptoms
* Already included in PFBIO or included simultaneously in PFBIO and PFBIO-EXA
* Age at least 18 years

Exclusion Criteria:

* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients already included in PFBIO that are admitted with a respiratory worsening are eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-06-13 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
  All-cause mortality
Mortality | 90 days
  All-cause mortality

SECONDARY OUTCOMES:
Biomarker levels | 30 days
  Blood biomarker level
LTOT | 30 days
  Change in oxygen need
QoL | 30 days
  Score of patient reported quality of life assessed by questionnaires
Respiratory support | 30 days
  Need for non-invasive or invasive respiratory support, including oxygen, CPAP, NIV and intubation
Decline in functional level | 30 days
  Decrease in functional level, e.g. moved to nursing home, hospice or other
Treatment during hospitalization | 30 days
  Treatment administered for respiratory worsening
Treatment after hospitalization | 90 days
  Treatment administered after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev and Gentofte Hospital, Hellerup, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No